CLINICAL TRIAL: NCT02994940
Title: Modified Pre-operative Oral Doses Acetaminophen Versus Intravenous Acetaminophen
Acronym: MODIV-APAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 948256
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Tonsillectomy; Adenoidectomy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Acetaminophen (Experimental): Group 1 will receive oral acetaminophen 30mg/kg 30-60 minutes prior to scheduled surgery time . Group 1 patients will receive placebo IV infusion just prior to surgery incision.
  Interventions: Drug: Acetaminophen
- Intravenous Acetaminophen (Experimental): Group 2 will receive placebo oral medication at approximately 30-60 minutes prior to scheduled surgery. Group 2 patients will receive IV acetaminophen 15 mg/kg just prior to surgery incision.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — already included in arm/group descriptions
  Other Names: OFIRMEV

SUMMARY:
Acetaminophen is frequently used as an adjunct for pain management in pediatric surgical patients. The drug is available in an over the counter, inexpensive oral form as well as a considerably more expensive intravenous form. This study will compare opioid requirements and acetaminophen plasma levels post operatively for two dosing regimens to compare oral versus intravenous routes given pre operatively.

DETAILED DESCRIPTION:
The primary purpose of this study is to compare opioid utilization in post-operative patients undergoing tonsillectomy and adenoidectomy, between IV and PO acetaminophen. Secondarily, it will provide information regarding possible cost savings, pharmacokinetics and safety between these two regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 3 years to 17 years scheduled for tonsillectomy and adenoidectomy for obstructive sleep apnea with or without additional minor procedures such as sleep endoscopy, unilateral or bilateral myringotomy, insertion of tympanostomy tubes and/or ear exam. ( Minor additional procedures that are frequently combined with tonsillectomy and adenoidectomy but are not commonly considered to have pain that is significantly greater than the tonsillectomy and adenoidectomy).

Exclusion Criteria:

* Patients who meet University of California Davis Children's Hospital (UCDCH) criteria for Pediatric Intensive Care Unit (PICU) admission: on home oxygen pre-operatively, exhibit airway obstruction when awake (stertor above larynx, stridor at larynx), sleep study with apnea hypoxia index greater than 25 or sleep oxygen saturation nadir <80%, cardiac disease, difficult intubation.
* Patients with a known allergy to acetaminophen
* Patients with known hepatic insufficiency or severe hepatic disease
* Patients with known Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients who are malnourished (ie lower levels of glutathione)
* Patients with severe renal impairment as defined by calculated creatinine clearance <20 ml/min (per modified Schwarz equation)
* Patients who are pregnant

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Lammers, MD, Principal Investigator — UC Davis Children's Hospital
Locations (1):
- University of California Davis Children's Hospital, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lammers CR, Schwinghammer AJ, Hall B, Kriss RS, Aizenberg DA, Funamura JL, Senders CW, Nittur V, Applegate RL 2nd. Comparison of Oral Loading Dose to Intravenous Acetaminophen in Children for Analgesia After Tonsillectomy and Adenoidectomy: A Randomized Clinical Trial. Anesth Analg. 2021 Dec 1;133(6):1568-1576. doi: 10.1213/ANE.0000000000005678. PMID 34304234

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Acetaminophen: Group 1 will receive oral acetaminophen 30mg/kg 30-60 minutes prior to scheduled surgery time . Group 1 patients will receive placebo IV infusion just prior to surgery incision.
  Acetaminophen
- Intravenous Acetaminophen: Group 2 will receive placebo oral medication at approximately 30-60 minutes prior to scheduled surgery. Group 2 patients will receive IV acetaminophen 15 mg/kg just prior to surgery incision.
  Acetaminophen
Period: Overall Study
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Started | 37 | 37
Completed | 30 | 36
Not Completed | 7 | 1
Not completed — Did not receive study medications: Study drug not available prior to anesthesia induction | 6 | 0
Not completed — Did not receive study medications: vomited after ingestion | 1 | 0
Not completed — Did not receive study medications: red dye allergy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Completed subjects (n=66) used for analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen | Total
Number analyzed (Participants) | 30 | 36 | 66
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4 [4 to 8] | 6 [4.3 to 7] | 5 [4 to 7.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 15 | 22 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 19.3 [16.6 to 25.3] | 20.6 [18.3 to 28.2] | 20.2 [17.5 to 25.7]
Percentile weight for age [Median (Inter-Quartile Range); unit: percentile] | 55.0 [27.0 to 86.3] | 45.0 [29.3 to 84.8] | 49.5 [29.8 to 85.5]

OUTCOME MEASURES:

1. Primary Outcome: Total Dose of Opioid
Description: Total dose of opioid, in morphine equivalents, that the patient receives for breakthrough pain in the 24 hour period following surgery.
Time Frame: Within 24hrs
Measure: Median (Inter-Quartile Range); unit: mcg/kg
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 30 | 36
mcg/kg | 147.6 [119.6 to 193.0] | 125.4 [102.8 to 150.9]
Statistical Analysis 1: Comparison: Oral Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.127, Wilcoxon (Mann-Whitney); Hodges Lehman estimator = 21.3, 95% CI 2-sided [-2.5 to 44.2]

2. Secondary Outcome: Proportion of Patients With Severe Pain Score of 7 or Higher
Description: A secondary endpoint is the proportion of patients with pain scores in the severe pain range (7 or higher) on numeric pain rating scale of 0 to 10; higher score more severe.
Time Frame: 24 hrs period following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 30 | 36
Participants | 15 | 17
Statistical Analysis 1: Comparison: Oral Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.851, Chi-squared

3. Secondary Outcome: Plasma Acetaminophen Level 1 - End of Surgery
Description: mg/L acetaminophen in the plasma at the end of surgery
Time Frame: at the end of surgery, about 1 hour after IV Dose
Population: 2 patients in Oral did not have sample obtained for level; 1 patient in IV had value below 10 mg/L limit of quantification
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 28 | 35
mg/L | 22 [16.5 to 27.8] | 20 [17 to 22]
Statistical Analysis 1: Comparison: Oral Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.109, Wilcoxon (Mann-Whitney); Hodges Lehman estimator = 2.0, 95% CI 2-sided [-1.0 to 6.0]

4. Secondary Outcome: Plasma Acetaminophen Level 2 - 3 Hours After IV Study Drug Administration
Description: mg/L acetaminophen in the plasma 3 hours after IV study drug administration
Time Frame: Outcome will be measured 3hrs post first IV Dose
Population: Acetaminophen plasma levels obtained 3 hours after start of the IV study drug in patients with samples obtained; these were not available for 8 Oral and 9 IV subjects.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 21 | 16
mg/L | 18 [15.0 to 21.0] | 11 [10.3 to 12.8]
Statistical Analysis 1: Comparison: Oral Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney); Hodges Lehman estimator = 7.0, 95% CI 2-sided [4.0 to 8.0]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Oral Acetaminophen | Intravenous Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/36
Other Adverse Events (participants affected / at risk) | 0/30 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT02994940/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT02994940/ICF_001.pdf